CLINICAL TRIAL: NCT00836758
Title: Validation of Breathing Event Detection of the REMstar Auto With Aflex Compared to Clinical Polysomnography
Brief Title: Comparison of Breathing Event Detection by a Continuous Positive Airway Pressure Device to Clinical Polysomnography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDILP-2008-SST-01
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-12

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Participants wore a PAP device and had a PSG at the same time. These participants had their PSG data compared to the PAP data.
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP Device (Experimental): Breathing event detection (AED) by the CPAP device will be compared to breathing event detection by a simultaneous PSG (manual PSG scoring).
  Interventions: Device: Analysis with AED and manual PSG scoring

INTERVENTIONS:
Device: Analysis with AED and manual PSG scoring — The CPAP device will be set-up at a sub-therapeutic pressure and will remain at this pressure for the entire night, if tolerated. Then the events will be analyzed with Automatic Event Detection (AED) and manual PSG scoring.

SUMMARY:
The study is to compare the performance of a CPAP (continuous positive airway pressure) device to a clinical polysomnography (PSG) in identifying breathing events in patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
Purpose: The purpose of this study was to compare the AED algorithm used in a PAP device with manually scored events on PSG. The PAP device was modified to produce a square wave voltage output identifying when apneas, hypopneas, and snoring events were detected. Recording this event signal on the PSG performed with the patient using the PAP device allowed an event-by-event comparison between manually scored PSG events and AED events. In addition, the AHI, AI, and HI derived from the manually scored PSG were compared with the respective measures reported by the PAP device used during the PSG.

Study Objectives: Compare automatic event detection (AED) of respiratory events using a positive airway pressure (PAP) device with manual scoring of polysomnography (PSG) during PAP treatment of obstructive sleep apnea (OSA).

Design: Prospective PSGs of patients using a PAP device.

Setting: Six academic and private sleep disorders centers.

Interventions: A signal generated by the PAP device identifying the AED of respiratory events based on airflow was recorded during PSG.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-75
2. Diagnosis of OSAHS with a baseline AHI ≥ 15 events/hr of sleep assessed January 01, 2007 or later
3. CPAP prescription of 8cm of H20 or higher
4. Able and willing to provide written informed consent
5. Native English speaker

Exclusion Criteria:

1. Participation in another interventional research study within the last 30 days
2. Major medical or psychiatric condition that would interfere with the demands of the study and adherence to PAP. Examples include unstable cardiovascular disease (Class III / IV CHF), neuromuscular disease, cancer, and renal failure.
3. Chronic respiratory failure or insufficiency with suspected or known neuromuscular disease, moderate or severe continuous positive airway pressure (COPD) or other pulmonary disorders, or any condition with an elevation of arterial carbon dioxide levels (> 45 mmHg) while awake, or subjects requiring continuous oxygen therapy.
4. Surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days
5. Surgery at any time for the treatment of OSAHS such as uvulopalatopharyngoplasty (UPPP)
6. Presence of untreated or poorly managed,non-OSAHS related sleep disorders:

   1. moderate to severe periodic limb movements(≥ 30/hr with symptoms or arousals)
   2. arousals associated with periodic limb movements > 10 per hour or
   3. anyone experiencing chronic and severe insomnia.
7. Consumption of ethanol immediately prior to the research PSG

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Berry, MD, Principal Investigator — University of Florida
Locations (1):
- Shands and UF Sleep Disorder Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 148 (PSGs and overnights with PAP therapy), collected from 115 unique participants, were included in this analysis.
Pre-assignment Details: 119 studies had a technically adequate recording and were collected from 90 patients (29 patients participated in two studies).
  These 119 studies were pooled with another 29 studies from another trial for a total of 148 studies. 4 patients participated in both trials and 3 of these patients contributed two recordings.
Units Other Than Participants: Overnight PSG and AED algorithms
Groups:
- All Participants: Data was collected from participants that participated in a multi-center, randomized, double-blind trial comparing three modes of positive pressure delivery who had overnight PSGs.
Period: Overall Study
Arm/Group | All Participants
Started | 115; 148 Overnight PSG and AED algorithms
Completed | 115; 148 Overnight PSG and AED algorithms
Not Completed | 0; 0 Overnight PSG and AED algorithms

BASELINE CHARACTERISTICS:
Population: *In summarizing the age, BMI, and sex statistics, the 4 participants who completed both trials were only counted once.
Groups:
- CPAP Device: Breathing event detection (AED) by the continuous positive airway pressure (CPAP) device will be compared to breathing event detection by a simultaneous PSG (manual PSG scoring).
  Analysis with AED and manual PSG scoring: The CPAP device will be set-up at a sub-therapeutic pressure and will remain at this pressure for the entire night, if tolerated. Then the events will be analyzed with Automatic Event Detection (AED) and manual PSG scoring.
Arm/Group | CPAP Device
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 84
Region of Enrollment [Number; unit: participants]
  United States | 115
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.2 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Indices (AHI) as Determined by Polysomnography (PSG) vs Automatic Event Detection (AED ) Algorithm
Description: Apnea-hypopnea index (AHI) is the combined average number of apneas and hypopneas that occur per hour of sleep. The Apnea index (AI) is the average number of apneas that occur per hour of sleep. The Hypopnea index (HI) is the average number of hypopneas that occur per hour of sleep.
  The PSGs were manually scored to determine the apnea-hypopnea index. This value was then compared to the PAP device which utilized the AED algorithm to determine the apnea-hypopnea index.
Time Frame: one night
Measure: Mean (Standard Deviation); unit: events per hour
Units Other Than Participants: Overnight PSG and AED algorithms
Groups:
- Manual PSG Scoring: The PSGs were manually scored with the aid of computer software by a PSG technologist at a central scoring facility. The technologist was blinded to the event signal during manual scoring (the event signal was not visible in the montages used for scoring). Sleep staging and respiratory events were scored using 2007 American Academy of Sleep Medicine (AASM) guidelines. The scoring of a hypopnea required that the event be associated with a ≥ 4% oxygen desaturation.
- Automatic Event Detection: The AED algorithm used the following criteria to identify respiratory events. An apnea was detected when there was an 80% or greater reduction in the airflow for 10 sec or longer in comparison with the average airflow over the previous 2 minutes. A hypopnea was detected when there was a device estimated 40% reduction in airflow for ≥ 10 sec but < 60 sec compared with the average airflow over the previous 2 minutes. The hypopnea detection algorithm required the presence of two recovery breaths that nominally were at least 75% to 80% of the baseline airflow. The algorithm also looked for evidence of flow limitation to detect hypopneas. The algorithm monitored the flow signal for changes in peak flow, and the shape of the inspiratory airflow signal that would be associated with flow limited breathing.
Arm/Group | Manual PSG Scoring | Automatic Event Detection
Number analyzed (Participants) | 115 | 115
Number analyzed (Overnight PSG and AED algorithms) | 148 | 148
events per hour
  Apnea-hypopnea index | 5.6 (8.0) | 5.8 (6.3)
  Apnea index | 2.4 (4.8) | 3.2 (5.25)
  Hypopnea index | 3.2 (5.2) | 2.6 (2.3)
Statistical Analysis 1: Comparison: Manual PSG Scoring vs Automatic Event Detection; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Methodological Comparisons of AHI, Apnea Index (AI) and Hypopnea Index (HI) as Determined by Intra-class Correlation (ICC)
Description: Methodological comparisons utilizing ICC for detection of AHI, apnea index (AI) and hypopnea index (HI) were caculated between the values obtained by PSG and the REMstar Auto with A-Flex device.
Time Frame: one night
Measure: Number; unit: coefficient
Units Other Than Participants: Overnight PSG and AED algorithms
Groups:
- CPAP Device Compared to Manual PSG Scoring: This analysis focused on events detected by the CPAP device compared to Manual PSG scoring. The two arms were compared to demonstrate agreement.
Arm/Group | CPAP Device Compared to Manual PSG Scoring
Number analyzed (Participants) | 115
Number analyzed (Overnight PSG and AED algorithms) | 148
coefficient
  Apnea-Hypopnea Index | 0.789
  Apnea Index | 0.825
  Hypopnea Index | 0.350

ADVERSE EVENTS:
Time Frame: one overnight visit
Description: As this was a review of overnight data from another study, there were no adverse events or serious adverse events, as only data was reviewed.
Arm/Group | CPAP Device
All-Cause Mortality (participants affected / at risk) | 0/115
Serious Adverse Events (participants affected / at risk) | 0/115
Other Adverse Events (participants affected / at risk) | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No